CLINICAL TRIAL: NCT04943016
Title: Phase I Clinical Trial of CD19 Chimeric Antigen Receptor (CAR) T Cells in Children and Adults With Relapsed or Refractory CD19 Positive B Cell Malignancies
Brief Title: CD19 CAR T Cells in Children and Adults With Relapsed or Refractory CD19 Positive B Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202103150MINC
Record Dates: First submitted 2021-06-04; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-05

CONDITIONS: Relapsed/Refractory B-Cell Malignancies
MeSH Terms: conditions — Recurrence | interventions — Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 Chimeric Antigen Receptor (CAR) T Cells (Experimental): The dose is escalated in standard 3 +3 design with a starting dose of 1x10^6 cell/kilogram and maximum treatment dose of 5 x 10^6 cell/kilogram. The minimum number of 9 subjects would occur if no dose-limiting toxicities are observed in the 3 dose escalation cohorts. The maximum sample size of 18 subjects would be enrolled in 3 dose escalation cohorts (six in each cohort) for meeting dose-limiting toxicities request. In addition, we hypothesize that we will be able to successfully manufacture CAR T cells to meet the established release criteria at a minimum target dose of 1 X 106 +-30% cells/kilogram in this patient population using the Miltenyi CliniMACS Prodigy® closed transduction system.
  Interventions: Drug: CD19 Chimeric Antigen Receptor (CAR) T Cells

INTERVENTIONS:
Drug: CD19 Chimeric Antigen Receptor (CAR) T Cells — This study seeks to examine the feasibility and safety of the administration of autologous T cells that have been modified through the introduction of a chimeric antigen receptor targeting the B cell surface antigen CD19 following administration of chemotherapy lymphodepletion regimen in children and adults with relapsed/refractory B cell malignancies. The overall goal of this study is to validate the safety profile of administration CD19 CAR T cells and describe the toxicities in children and adults with relapsed/ refractory B cell malignancies. Each patient implements leukapheresis 2 weeks after enrollment and infuse CD19 CAR-T cell around 2 weeks after leukapheresis, and administrated chemotherapy lymphodepletion regimen 1 week before infusion. Furthermore, the treated subject would be following up around 2 years.

SUMMARY:
This study seeks to examine the feasibility and safety of the administration of autologous T cells that have been modified through the introduction of a chimeric antigen receptor targeting the B cell surface antigen CD19 following administration of chemotherapy lymphodepletion regimen in children and adults with relapsed/refractory B cell malignancies.

DETAILED DESCRIPTION:
The overall goal of this study is to validate the safety profile of administration CD19 CAR T cells and describe the toxicities in children and adults with relapsed/ refractory B cell malignancies. The dose is escalated in standard 3 +3 design with a starting dose of

1x106 cell/kilogram and maximum treatment dose of 5 x 106 cell/kilogram. The minimum number of 9 subjects would occur if no dose-limiting toxicities are observed in the 3 dose escalation cohorts. The maximum sample size of 18 subjects would be enrolled in 3 dose escalation cohorts (six in each cohort) for meeting dose-limiting toxicities request. In addition, we hypothesize that we will be able to successfully manufacture CAR T cells to meet the established release criteria at a minimum target dose of 1 X 106 +-30% cells/kilogram in this patient population using the Miltenyi CliniMACS Prodigy® closed transduction system.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have the ability to understand and the willingness to sign a written informed consent document
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, between the age of 1 and 65 years
4. In good general health as evidenced by medical history and diagnosed relapsed or refractory CD19+ B cell malignancies including acute lymphocytic leukemia (ALL), non-Hodgkin's lymphoma containing Diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL), follicular lymphoma (FL), or small lymphocytic lymphoma (SLL), B-cell prolymphocytic leukemia(BPLL), Lymphoplasmacytic Lymphoma, Marginal Zone Lymphoma (MZL).
5. Definition of relapse or refractory as below:

   * Ineligible hematopoietic transplantation
   * Relapse after transplantation
   * Subject with ALL was evaluated by minimal residual disease > 0.1% after treatment with at least two lines of therapy. Subjects with Philadelphia Chromosome positive acute lymphoblastic leukemia (Ph+ALL) treated by at least two lines of therapy, including tyrosine kinase inhibitors (TKIs) are eligible.
   * Subject with lymphoma treated regimens containing both anti-CD20 antibody and anthracycline-containing chemotherapy regiment. Subjects with transformed follicular lymphoma must have received prior chemotherapy for follicular lymphoma and subsequently have the chemo refractory disease after transformation to diffuse large B-cell lymphoma
6. The patient's disease must be CD19 positive, either by immunohistochemistry or flow cytometry analysis on the last biopsy available.
7. Performance status: Adult Subjects: ECOG ≤2; Subjects > 10 years of age: Karnofsky≥ 50%; Subjects ≤ 10 years of age: Lansky scale ≥ 50% (See Appendix 1)
8. The following laboratory values :

   * Total bilirubin ≤ 2x upper limit of normal
   * AST (SGOT) ≤ 5x upper limit of normal
   * ALT (SGPT) ≤ 5x upper limit of normal
   * Serum Creatinine ≤ 2.0 mg/dl
   * Subjects must have the following hematologic function parameters (supportive care is allowed per institutional standards, i.e. filgrastim, transfusion):

     i.Absolute lymphocyte count>0.3× 109cells/L ii.Platelets>50 × 109 cells/L
9. Prior therapy wash-out: At least 2 weeks or 5 half-lives, whichever is longer, must have elapsed since any prior systemic therapy including cytotoxic chemotherapy, immunomodulatory, immunosuppressive, antiproliferative drugs, antibody, immune checkpoint therapy, pegylatedasparaginase, pegfilgrastimat the time the subject is planned for leukapheresis. Filgrastim, intrathecal methotrexate, systemic steroid, and donor lymphocyte infusion must be stopped 5 days, 7 days, 72 hours, and 4 weeks before leukapheresis, respectively.
10. Ability to take oral medication and be willing to adhere to the intervention protocols and medication regimens
11. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during the follow-up period of the protocol
12. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

1. Current use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary.
2. Pregnancy or lactation
3. Known allergic reactions to components used in the intervention protocols or medication regimens in this study
4. Active Febrile illness
5. Treatment with another investigational drug or other intervention within 30 days or 5 half-lives.
6. Autologous transplant within 6weeks of planned CAR-T cell infusion.
7. Patients who are able to obtain market approved CD19 CAR T-cell therapies.
8. Active central nervous system or meningeal involvement by tumor. Subjects with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of CNS or meningeal involvement must be in a documented remission by CSF evaluation and contrast-enhanced MRI imaging for at least 90 days prior to Enrollment.
9. History of active malignancy other than non-melanoma skin cancer, carcinoma in situ (e.g. cervix, bladder, breast).
10. Active HIV infection.
11. Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
12. Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of child-bearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study to the follow-up period of the protocol.
13. Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
14. Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative viral load prior to enrollment. (viral load positive patients will be excluded.)
15. Severe concomitant disease or organic dysfunction that is expected to reduce life expectancy less than 3 months.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
80% Proportion of products successfully manufactured meeting the established release criteria with a goal of at least CAR-T cell 1 X 10^6 cells/kilogram. | 3 years
  To examine the feasibility of manufacture of autologous CD19 CAR T-cells at a minimum target dose of 1 X 106 cells/kilogram using the Miltenyi CliniMACS Prodigy® automated system
Incidence and severity of adverse events | 3 years
  To determine the safety of infusion with chimeric antigen receptor T cells targeting CD19
Incidence and severity of Dose Limited Toxicities | 3 years
  Find the recommended phase II dose (RP2D) for recurrent/refractory B cell malignancies
Incidence and severity of Maximum Toxicity Dose | 3 year
  Find the recommended phase II dose (RP2D) for recurrent/refractory B cell malignancies

IPD SHARING:
Plan to Share IPD: No